CLINICAL TRIAL: NCT04336865
Title: Effect of Hormonal Contraception on Lower Urinary Tract Symptoms& Sexual Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, randa habeeb yacoup, resident doctor, Assiut University
Other Study IDs: hormonal contraception
Record Dates: First submitted 2020-04-04; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Effect of hormonal contraception on lower urinary tract symptoms& sexual function

DETAILED DESCRIPTION:
It is generally accepted that female sex hormones influence the morphology and physiology of vaginal tissues. Peripheral estrogen affects urogenital connective tissue composition and structure, vaginal blood flow, and thickness of vaginal epithelium. Estrogen and progestagen receptors are also abundantly present in the lower urinary tract, which has the same embryonic origin as the vagina. decline in circulating estrogen levels may result in atrophy of vaginal, urethral and bladder trigonal epithelium, as well as initiate metabolic changes in the subepithelial supportive tissues. This process forms the biological rationale for the common clinical practice of prescribing hormone treatment to menopausal women with lower urinary and genital tract symptoms.

Contrary to widespread belief, the Womens Health Initiative (WHI) randomised trial showed that menopausal hormone therapy with conjugated estrogen alone, or in combination with progestagen, increased the risk of de novo or aggravated urinary incontinence after one year of treatment. In premenopausal women, oral contraception is the most common source of hormone intake but very few studies have endeavored to determine the effects of oral contraception on premenopausal urinary incontinence. The aim of this nationwide cohort study was to assess the influence of contraceptives on the risk for lower urinary tract dysfunction in young female.at is time-related with the beginning of hormonal contraception, health care providers should give information about other methods and try to switch them to a method less associated with sexual dysfunction. However, there are contradictory results between the different studies regarding the association between sexual dysfunction and hormonal contraceptives, so it could be firmly said that additional research is needed.

Meanwhile, it could be said that hormonal contraception has been associated with different alterations in sexual functioning.

To conclude, a multidisciplinary approach to the management of female sexual dysfunction is mandatory, and health care providers should give lifestyle counselling apart from proposing different treatment options. An adequate relationship with the patient, as well as the routine monitoring of possible sexual dysfunction, are essential in addressing these difficulties. Undoubtedly, the best contraceptive is one that fulfills the women's needs with acceptable side effects and agreed with the prescribed

ELIGIBILITY:
Inclusion Criteria:

1. Women taking hormonal contraception e.g cocs .pops.implanon&.injectable contraception
2. Women has good regular marital life

Exclusion Criteria:

1. female has organic urinary dysfunction
2. female has mental& psycological dysfunction
3. chronic disease DM.hypertension. chronic renal disease
4. prolapse
5. previous perineal &vaginal correlation surgery
6. women taking any treatment for urinary tract infection &sexual dysfunction

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: all women attending family planning clinic taking hormonal contraception
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Arabic female sexual function index | baseline
  valid questionnaire that can be used in the Egyptian population. The questionnaire is relatively easy to be understood by lay women and does not contain unacceptably sexually explicit questions, which may pose difﬁculties for self-rating. ArFSf I is valid and reliable,and it is as good as the original FSFI in assessing female sexual function &good psychometric tool for sexual dysfunction . Research in the area of female sexuality is not easy and relatively challenging in the Arab world
Bristol female lower urinary tract symptoms questionnaire | baseline
  it was designed to asses lower urinary tract symptoms in women & quality of sexual life . it will be translated into arabic language

CONTACTS AND LOCATIONS:
Overall Officials: muhmoud zakhera, Study Chair — Assiut University; mostafa bahlool, Study Chair — Assiut University
Locations (1):
- Women"S Health Hospital, Asyut, Egypt

REFERENCES:
- [Background] Batra SC, Iosif CS. Progesterone receptors in the female lower urinary tract. J Urol. 1987 Nov;138(5):1301-4. doi: 10.1016/s0022-5347(17)43588-9. PMID 3669191
- [Background] Champaneria R, D'Andrea RM, Latthe PM. Hormonal contraception and pelvic floor function: a systematic review. Int Urogynecol J. 2016 May;27(5):709-22. doi: 10.1007/s00192-015-2833-3. Epub 2015 Sep 25. PMID 26407563
- [Background] de Castro Coelho F, Barros C. The Potential of Hormonal Contraception to Influence Female Sexuality. Int J Reprod Med. 2019 Mar 3;2019:9701384. doi: 10.1155/2019/9701384. eCollection 2019. PMID 30941356